CLINICAL TRIAL: NCT06842134
Title: Phase 1, Prospective, Single-Center, Randomized Sequence, Open Label, 2-Way Crossover Study Comparing Organic Phosphate (Sodium Glycerophosphate Injection) to Numeta G16%E.
Brief Title: A Study Comparing Organic Phosphate (Sodium Glycerophosphate Injection) to Numeta G16%E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BXU561373 (B)
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Parenteral Nutrition
Keywords: organic phosphate; inorganic phosphate; sodium glycerophosphate; pharmacokinetic; intravenous; parenteral nutrition
MeSH Terms: conditions — Hyperphagia | interventions — alpha-glycerophosphoric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence CD (Numeta G16%E/Organic phosphate) (Experimental): * Period 1: Regimen C (Numeta G16%E)
  * Period 2: Regimen D (Organic phosphate (sodium glycerophosphate SGP))
  Interventions: Drug: Numeta G16%E; Drug: Sodium Glycerophosphate Injection
- Sequence DC (Organic phosphate/Numeta G16%E) (Experimental): * Period 1: Regimen D (Organic phosphate (sodium glycerophosphate SGP))
  * Period 2: Regimen C (Numeta G16%E)
  Interventions: Drug: Numeta G16%E; Drug: Sodium Glycerophosphate Injection

INTERVENTIONS:
Drug: Numeta G16%E — Numeta G16%E (1000mL) will be given intravenously via peripherally inserted central catheter and will provide an equimolar IV phosphate dose of 8.7 mmol over 9 h.
Drug: Sodium Glycerophosphate Injection — Organic phosphate (SGP) will be diluted 1000mL of sodium chloride (0.9% normal saline) to achieve an equimolar IV phosphate dose of 8.7 mmol over 9 h.

SUMMARY:
This is a phase 1, prospective, single-center, randomized sequence, open label, 2-way crossover study comparing Organic Phosphate (Sodium Glycerophosphate Injection) to Numeta G16%E.

It is planned to randomize approximately 16 healthy male and female subjects. All study periods will be completed during a single residency, the overall duration of residency will be 11 days (10 nights).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females.
2. Aged 18 to 55 years, inclusive, at the time of signing informed consent.
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 and a minimum body weight of 57 kg as measured at screening.
4. Must be willing and able to comply with all study requirements including dietary requirements.
5. Subject must be literate, has signed a written informed consent form (ICF) and has the ability to communicate and comply with all study requirements
6. Must agree to use an adequate method of contraception.
7. Alkaline phosphatase level within standard reference range/normal limits at screening and admission.
8. Serum inorganic phosphate level within standard reference range/normal limits at screening and admission.
9. Serum parathyroid hormone (PTH) level within standard reference range/normal limits at screening.
10. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels within reference range/normal limits at screening and admission.

Exclusion Criteria:

1. Subjects who have received any investigational medicinal product (IMP) in a clinical research study within 5 half-lives or within 30 days prior to first dose, whichever is longer.
2. Subjects who are study site or Sponsor employees, or subjects who are immediate family members of study site or Sponsor employees.
3. Subjects who have previously been administered IMP in this study.
4. History of any drug or alcohol abuse in the past 2 years prior to screening.
5. Regular alcohol consumption in 6 months prior to screening.
6. A confirmed positive alcohol urine test at screening or admission.
7. Current smokers or those who have smoked within the last 12 months prior to screening. A confirmed positive urine cotinine test at screening or first admission.
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months prior to screening.
9. Females of childbearing potential must have a negative pregnancy test (urine pregnancy test at screening). Females who are pregnant or lactating will be excluded.
10. Have poor venous access that limits phlebotomy.
11. Clinically significant abnormal clinical chemistry or hematology as judged by the Investigator.
12. Clinically significant abnormal urinalysis as judged by the Investigator.
13. History of diabetes mellitus (types I or II).
14. Prediabetes (fasting blood sugar level of >106 (repeat x 1 for confirmation of abnormal level).
15. Hypertriglyceridemia (fasting triglyceride level of > 200 mg/dL) at screening.
16. Subjects who, in the Investigator's opinion, have a clinically significant abnormal 12-lead resting ECG.
17. Positive drugs of abuse test result.
18. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
19. Evidence of renal impairment at screening, as indicated by an eGFR < 90mL/min/m^2.
20. History of any active systemic or immunologic disease, including but not limited to active renal, hepatic, hematological, gastrointestinal (except appendectomies/cholecystectomy), endocrinal, pulmonary (including asthma), cardiovascular, neurologic, or neurological disease (including demyelinating diseases such as multiple sclerosis), hypertension, tuberculosis, or systemic fungal infection.
21. History of bleeding ulcer, bleeding abnormalities or coagulation abnormalities.
22. History of hypophosphatasia.
23. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
24. Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator. Hay fever is allowed unless it is active.
25. Significant serious active skin disease, including rash, food allergy, eczema, psoriasis, or urticaria.
26. Donation or loss of 1 pint of blood within 3 months, or donation of plasma within 7 days prior to first dose of study medication or had a transfusion of any blood product within 3 months prior to study drug administration.
27. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g per day acetaminophen and HRT/hormonal contraception) within the last 30 days or five half-lives (whichever is longer), before IMP administration. Exceptions may apply on a case-by-case basis, if considered not to interfere with the objectives of the study, as determined by the Investigator.
28. Subjects who have been administered a drug by depot injection within 30 days prior to the initial study drug administration or 6 half-lives of that drug, whichever is longer and at the discretion of the Investigator or who have received a recent (as determined by the Investigator) live or attenuated vaccination (with exception of a COVID-19 vaccine or flu vaccine), or exposure to communicable viral diseases such as chicken pox, varicella, and measles.
29. Failure to satisfy the Investigator of fitness to participate for any other reason.
30. Known hypersensitivity to egg, soya or peanut proteins.
31. Food allergies deemed clinically relevant by the investigator which would hinder ability to adhere to the prescribed diet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Baseline-corrected maximum observed concentration (C(maxbc)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Baseline-corrected area under the curve from time 0 to 24h post-dose (AUC(0-24bc)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter

SECONDARY OUTCOMES:
Baseline-corrected total urinary inorganic phosphate excreted in the urine (Ae(0-24bc)) | Days 1 and 7
  Urine PK parameter
Time of maximum observed concentration (T(max)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Apparent terminal elimination half-life (T(1/2 z)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Elimination rate constant (K(z)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Maximum observed concentration (C(max)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Area under the curve from time 0 to 24h post-dose (AUC(0-24)) for inorganic phosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Total urinary inorganic phosphate excreted in the urine (Ae(0-24)) | Days 1 and 7
  Urine PK parameter
Baseline-corrected time of maximum observed concentration (T(maxbc)) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
T(max) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Baseline-corrected apparent terminal elimination half-life (T(1/2 zbc)) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
T(1/2 z) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
Baseline-corrected elimination rate constant (K(zbc)) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
K(z) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
C(maxbc) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
C(max) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
AUC(0-24bc) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
AUC(0-24) for glycerophosphate | Days 1, 2, 7, and 8
  Serum PK parameter
T(maxbc) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
T(max) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
T(1/2 zbc) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
T(1/2 z) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
K(zbc) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
K(z) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
C(maxbc) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
C(max) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
AUC(0-24bc) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
AUC(0-24) for glycerol | Days 1, 2, 7, and 8
  Serum PK parameter
Change from baseline in Alanine Aminotransferase (ALT) | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in Alkaline Phosphatase | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in Aspartate Aminotransferase (AST) | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in total bilirubin | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in direct bilirubin | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in eGFR | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in Blood Urea Nitrogen (BUN) | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in creatinine | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in calcium | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in phosphate | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in magnesium | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in potassium | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in sodium | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in respiratory rate | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in heart rate | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in temperature | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Change from baseline in blood pressure | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Number of subjects with any physical examination interpreted as abnormal | Baseline through Day 11
  Safety outcome
Number of subjects experiencing any clinically significant abnormality in ECGs | Baseline, Day 1, Day 2, Day 7, Day 8
  Safety outcome
Number of subjects experiencing adverse events | Baseline through Day 20
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Erika Ryan, DCN, MS, RD, CDN, CNSC, Study Director — Baxter Healthcare Corporation
Locations (1):
- Austin PPD CRU, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No